CLINICAL TRIAL: NCT02185261
Title: Interferon α for the Therapy of Minimal Residual Disease Following Hematopoietic Stem Cell Transplantation
Brief Title: Interferon α for the Therapy of Minimal Residual Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiaojun Huang, Peking University Institute of Hematology, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-02
Record Dates: First submitted 2014-02-10; First posted 2014-07-09 (Estimated); Last update posted 2018-06-07 (Actual); Status verified 2018-06

CONDITIONS: Leukemia
Keywords: Relapse; Minimal residual disease; Graft-versus-host disease; Acute leukemia; Interferon Alfa-2b
MeSH Terms: conditions — Leukemia; Recurrence; Neoplasm, Residual; Graft vs Host Disease | interventions — Interferon alpha-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- interferon Alfa-2b group (Experimental): Acute leukemia patients who are minimal residual disease positive after hematopoietic stem cell transplantation receive interferon Alfa-2b
  Interventions: Drug: Interferon Alfa-2b

INTERVENTIONS:
Drug: Interferon Alfa-2b — Patients who were deemed MRD-positive after day 60 post-transplantation receive interferon α-2b (subcutaneously at dosages of 3 million units 2-3 times per week) . Interferon treatment continues for 6 months in the absence of disease progression or unacceptable toxicity.
  Other Names: INF α-2b

SUMMARY:
This study aimed to evaluate the efficacy of interferon α among patients undergone unmanipulated blood and marrow transplantation following day 60 post-transplantation who were minimal residual disease positive after transplantation.

Hematopoietic stem cell transplantation (HSCT) is an effective treatment option for acute leukemia and many other hematological malignancies. However, post-transplant relapse can occur in some patients, and the prognosis of these patients is usually very poor.The persistence or recurrence of minimal residual disease (MRD) in the post-transplant period is an independent risk factor of relapse. Therefore, MRD monitoring can be used to screen patients with a high risk of relapse to provide timely intervention and prevent post-transplant relapse.Interferon α-2b exerts a relatively strong immunomodulatory effect. It can kill acute leukemia (AL) cells by regulating T-cell and/or natural killer cell functions.Consequently, interferon α-2b may have potential therapeutic value for AL patients with MRD-positive after transplantation.

The study hypothesis:

Prevention of relapse using interferon α-2b following hematopoietic stem cell transplantation in patients with standard risk acute leukemia can reduce relapse rate.

DETAILED DESCRIPTION:
Standard risk acute leukemia patients (except t(9;22)(q34; q11), t(15;17), inv(16)(p13q22), t(16;16)(p13; q22), or t(8;21)(q22; q22) cytogenetic abnormalities.) undergone unmanipulated blood and marrow transplantation following day 60 post-transplantation who were minimal residual disease positive after hematopoietic stem cell transplantation received interferon α-2b. The end points were safety and immunologic response. Following time is 12 months.

Primary Outcome Measures:

*The feasibility and efficacy of administering of subcutaneous interferon α-2b in this patient population. [ Time Frame: 1 years ]

Secondary Outcome Measures:

*The immunologic impact and clinical outcomes of subcutaneous interferon α-2b in patients after unmanipulated blood and marrow transplantation [ Time Frame: 1 years ] Estimated Enrollment:81 Study Start Date: Jun 2014 Estimated Study Completion Date: Jun 2016

Intervention Details Description:

*Drug:Interferon α-2b (subcutaneously at dosages of 3 million units 2-3 times per week) for 6 months in the absence of disease progression or unacceptable toxicity.

Acute leukemia patients who were MRD positive after day 60 post-transplantation receive interferon α-2b(subcutaneously at dosages of 3 million units 2-3 times per week). Interferon α-2b continues for 6 months in the absence of disease progression or unacceptable toxicity.

Participants will be seen periodically while they are receiving interferon α-2b. Physical exams and blood tests will be performed weekly for the first two weeks and then every other week until the completion of 6 months therapy.

Eligibility Ages Eligible for Study: 1-60 Years Genders Eligible for Study: Both Accepts Healthy Volunteers: No Criteria

The trial will be terminated in following situation

1. Severe toxicity occurrence
2. Cumulative incidence of relapse increased) (≥ 30%)
3. Cumulative incidence of mortality increased (≥ 30%)
4. Cumulative incidence of severe graft-versus-host disease increased (≥ 30%)
5. Although large enough sample had been enrolled, it did not reach statistical significance

ELIGIBILITY:
Inclusion Criteria:

* Patients who had standard-risk acute myeloid leukemia(CR1 or CR2) had minimal residual disease positive after hematopoietic stem cell transplantation

Exclusion Criteria:

* Patients with t(9;22)(q34; q11), t(15;17), inv(16)(p13q22), t(16;16)(p13; q22), or t(8;21)(q22; q22) cytogenetic abnormalities;active graft-versus-host disease; active infection; organ failure; exposure to donor lymphocyte infusion prior to enrollment

Ages: 1 Year to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 81 (Estimated)
Dates: Start 2014-06; Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
relapse rate | participants will be followed for an expected average of 1 year
  number of participants with morphologic relapse at one year

SECONDARY OUTCOMES:
The immunologic impact of subcutaneous interferon α-2b | participants will be followed for an expected average of 1 year
  examine the immune reconstitution of subgroups of T cells and nature killer cells after interferon α-2b application

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Jun Huang, MD, Principal Investigator — Peking University Institute of Hematology
Locations (1):
- Peking University Institute of Hematology,Beijing, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Shen MZ, Zhang XH, Xu LP, Wang Y, Yan CH, Chen H, Chen YH, Han W, Wang FR, Wang JZ, Zhao XS, Qin YZ, Chang YJ, Liu KY, Huang XJ, Mo XD. Preemptive Interferon-alpha Therapy Could Protect Against Relapse and Improve Survival of Acute Myeloid Leukemia Patients After Allogeneic Hematopoietic Stem Cell Transplantation: Long-Term Results of Two Registry Studies. Front Immunol. 2022 Jan 28;13:757002. doi: 10.3389/fimmu.2022.757002. eCollection 2022. PMID 35154096
- [Derived] Liu S, Luo X, Zhang X, Xu L, Wang Y, Yan C, Chen H, Chen Y, Han W, Wang F, Wang J, Liu K, Huang X, Mo X. Preemptive interferon-alpha treatment could protect against relapse and improve long-term survival of ALL patients after allo-HSCT. Sci Rep. 2020 Nov 19;10(1):20148. doi: 10.1038/s41598-020-77186-9. PMID 33214615
- [Derived] Chang YJ, Wang Y, Xu LP, Zhang XH, Chen H, Chen YH, Wang FR, Wei-Han, Sun YQ, Yan CH, Tang FF, Mo XD, Liu YR, Liu KY, Huang XJ. Haploidentical donor is preferred over matched sibling donor for pre-transplantation MRD positive ALL: a phase 3 genetically randomized study. J Hematol Oncol. 2020 Mar 30;13(1):27. doi: 10.1186/s13045-020-00860-y. PMID 32228710
- [Derived] Zhou YL, Wu LX, Peter Gale R, Wang ZL, Li JL, Jiang H, Jiang Q, Jiang B, Cao SB, Lou F, Sun Y, Wang CC, Liu YR, Wang Y, Chang YJ, Xu LP, Zhang XH, Liu KY, Ruan GR, Huang XJ. Mutation topography and risk stratification for de novo acute myeloid leukaemia with normal cytogenetics and no nucleophosmin 1 (NPM1) mutation or Fms-like tyrosine kinase 3 internal tandem duplication (FLT3-ITD). Br J Haematol. 2020 Jul;190(2):274-283. doi: 10.1111/bjh.16526. Epub 2020 Feb 26. PMID 32103499
- [Derived] Mo XD, Zhang XH, Xu LP, Wang Y, Yan CH, Chen H, Chen YH, Han W, Wang FR, Wang JZ, Liu KY, Huang XJ. IFN-alpha Is Effective for Treatment of Minimal Residual Disease in Patients with Acute Leukemia after Allogeneic Hematopoietic Stem Cell Transplantation: Results of a Registry Study. Biol Blood Marrow Transplant. 2017 Aug;23(8):1303-1310. doi: 10.1016/j.bbmt.2017.04.023. Epub 2017 Apr 27. PMID 28457953